CLINICAL TRIAL: NCT06764329
Title: The Effectiveness of Allogenic Mesenchymal Stem Cells Therapy on Hair Regrowth in Androgenetic Alopecia: a Randomized, Double-Blind, Placebo Control Trial
Brief Title: The Effectiveness of Allogenic Mesenchymal Stem Cells Therapy on Hair Regrowth in Androgenetic Alopecia.
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Collaborators: Pak Emirates Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFBMTC-2024-MSC in Alopecia
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Androgenetic Alopecia; Androgenetic Alopecia (AGA)
Keywords: androgenetic alopecia; mesenchymal stem cell; placebo-controlled trial
MeSH Terms: conditions — Alopecia | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo-Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): MSC therapy group
  Interventions: Biological: Mesenchymal Stem Cells
- Placebo group (Placebo Comparator): Placebo (0.9% saline)
  Interventions: Other: 0.9 % saline

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — allogeneic bone marrow-derived mesenchymal stem cells therapy
  Arms: Treatment
Other: 0.9 % saline — 0.9% Saline as placebo
  Arms: Placebo group

SUMMARY:
The goal of this study is to learn if mesenchymal stem cell therapy (treatment group) can effectively treat adrogenic alopecia or male-pattern baldness, when compared to normal saline (given to placebo group). It will also assess the differences in patient satisfaction. The main focus will be to:

1. Compare the average hair regenerative effect of mesenchymal stem cells versus Placebo, in treatment of androgenetic alopecia.
2. To determine and compare the investigators assessment and patient satisfaction in both groups.

Patients in treatment group will receive single session of MSC therapy injected in the scalp and placebo group will receive 0.9% saline solution. The participants will be followed for 12 weeks. The hair density and thickness will be mesured along with clinicians assessment and participant's satisfaction level.

DETAILED DESCRIPTION:
1. Introduction:

   Androgenetic Alopecia (AGA) is a common form of hair loss affecting both men and women, characterized by the miniaturization of hair follicles due to the influence of a variety of factors including androgens and genetics. AGA affects a sizeable portion of the population worldwide, affecting males and females both.1 While many accept it as a normal physiological process of ageing, for others it causes remarkable concern and worry, especially pertaining to personal appearance and self-confidence. So much so leading to body image issues and even psychological disorders1,2,3. Hence it becomes empirical to treat this condition with aim to achieve patient satisfaction. Current treatment options, such as minoxidil and finasteride, have limitations in efficacy and number of adverse effects which limit their use.1 Mesenchymal derived stem cells (MSCs) have emerged as a potential therapeutic option due to their regenerative and immunomodulatory properties.1 Cell-based therapy has seen a significant rise as an alternative for treating medical disorders in recent years. Specifically, stem cell therapy has been applied to address various dermatological conditions, including alopecia. Stem cells (SCs) are known to play a crucial role in initiating the hair growth cycle and remodeling.1 Emerging evidence suggests that stem cells may be responsible for releasing cytokines, chemokines, and specific growth factors like bFGF, VEGF, IGF-1, HGF, and TGF-β1. These molecules initiate cell repair processes through angiogenesis, immunomodulation, cell differentiation, and proliferation. In the scalp, they exert a paracrine effect on neighboring cells and tissues, promoting hair follicle growth, adjusting hair growth patterns, regulating follicle size via angiogenesis, and supporting the retention of the anagen phase.2,3 A RCT comparing Adipose derived Stem Cell Constituent Extract (ADSC-CE) with Placebo (Distilled water), carried out at Busan National University Yangsan Hospital, Korea showed significant statistical improvement in mean hair count and mean hair diameter in Intervention Group (IG) versus Control Group (CG) 16 weeks post treatment. Change from baseline in Hair Diameter was 0.008 ± 0.007 in IG versus 0.004 ± 0.004 in CG with p value of .023. Change from baseline in Hair counts was 3.89 ± 3.01 in IG versus 1.44 ± 1.97 in CG with p value of .025. In investigator assessment using photographs, intervention failed to show a statistically significant improvement in both groups. In the participants self-assessments, no significant intergroup differences were observed.3 Based on above evidence, there is a vast avenue of research in potential role of MSCs therapy in AGA, as an emerging approach.1,2,3 This study has the potential to pave the way for further advancements in regenerative medicine. This study aims to evaluate the efficacy and safety of MSCs in the treatment of AGA through a double-blind randomized controlled trial (RCT).

   As current treatments offer limited success, this study is directed to explore potential for a novel, minimally invasive alternative with long term effectiveness and improved outcomes in hair loss management, especially in our population, addressing an unmet clinical need.
2. OBJECTIVE i. To compare the mean hair regenerative effect of Mesenchymal derived stem cells (MSCs) versus Placebo, in treatment of androgenetic alopecia (AGA).

ii. To determine and compare the investigators assessment and patient satisfaction in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with AGA between age 25 to 59 years of age
* Clinical presentation consistent with Hamilton Norwood criteria grade ll to Vl
* Not currently receiving antiandrogens or minoxidil therapy.

Exclusion Criteria:

* Patients with hair loss other than AGA
* Patients receiving 5-alpha reductase inhibitor or minoxidil therapy
* Patients who received PRP for at least 6 months prior to enrollment
* History of hypertrophic scars or bleeding disorders
* History of treatment with hyper or hypothyroidism

Ages: 20 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in hair count | 12 weeks post intervention
  Primary efficacy variables will be the changes from baseline in hair count
Change in baseline hair diameter | 12 weeks post-intervention
  Change in baseline diameter measured through trichoscopic analysis.

SECONDARY OUTCOMES:
Investigators assessment through photographs of patients' scalp | 12 weeks post-intervention
  investigators assessment through photographs of patients' scalp pre- and post-intervention. An investigator, blinded to the intervention, will rate the changes in scalp appearance relative to the baseline using a standardized 7-point rating scale with the following scores:
  * 3 Greatly decreased
  * 2 Moderately decreased
  * 1 Slightly decreased 0 Unchanged
    * 1 Slightly increased
    * 2 Moderately increased
    * 3 Greatly increased
Subjective satisfaction of the patient | 12 weeks post-treatment
  Likert scale: subjective satisfaction of the patient, assessed through standardized questions regarding reduction in hair fall and new hair growth.
  Changes from baseline in terms of reduction in hairfall and new hair growth will be evaluated by the participants on a 5 point Likert Scale, post treatment (week 12).
  5. Extremely Dissatisfied 4. Satisfied 3. Neutral 2. Dissatisfied
  1. Extremely Dissatisfied

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Department of dermatology, Pak-Emirates Military Hospital, Rawalpindi
  - National Institute of Blood and Marrow Transplant (NIBMT), Rawalpindi

IPD SHARING:
Plan to Share IPD: No